CLINICAL TRIAL: NCT06552377
Title: A Cross-sectional Study Assessing the Agreement Between Sonographer Based Assessment of the Fatty Liver Using Conventional Ultrasound and Attenuation Imaging Scoring.
Brief Title: Ultrasound and Attenuation Imaging
Status: Completed | Type: Observational
Sponsor: Hywel Dda Health Board (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 329847
Record Dates: First submitted 2024-08-06; First posted 2024-08-14 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Fatty Liver; Non-alcoholic Steatohepatitis; Steatosis of Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All participants: Ultrasound attenuation imaging measurement
  Interventions: Device: Ultrasound Attenuation imaging measurement

INTERVENTIONS:
Device: Ultrasound Attenuation imaging measurement — Participant to undergo conventional ultrasound scanning with attenuation measurement as well.

SUMMARY:
Fatty liver disease affects almost a 3rd of the United Kingdom (UK) population. Currently, this is being investigated using a type of MRI scan that reports how fatty or not a person's liver is, with a liver fat score, but many patients cannot have this type of scan due to time, cost or because they have a condition which makes Magnetic Resonance Imaging (MRI) an unsafe scan for them to have. An ultrasound scan is cheaper, faster and safer for a wider variety of patients. New developments in ultrasound technology mean that instead of a Sonographer, or ultrasound operator, deciding whether your liver is fatty or not based on what they see on the scan, the ultrasound machine gives a liver fat score. This study will look at the relationship between the Sonographers' view on how fatty the liver is, compared with the liver fat score given by the new development in ultrasound technology.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) affects almost a 3rd of the population of the UK and current best practice is to evaluate this using Magnetic Resonance Imaging proton density fat fraction (MRI PDFF), however, this is inaccessible to many patients due to limited availability, cost and a large exclusion criteria. Ultrasound offers an affordable, faster and more inclusive method of liver evaluation but only subjective assessment of fatty liver disease until a recent development- Attenuation Imaging (AI). Attenuation imaging gives a numerical score for fatty liver disease. Attenuation imaging has previously only been compared to MRI PDFF, however, when many patients do not have MRI PDFF it is essential to compare it to common practice, conventional ultrasound. This study aims to assess the agreement between conventional ultrasound assessment of the liver and AI using a cross-sectional method. Convenience sampling will be used to select 95 participants who will have their AI score carried out alongside their routine ultrasound scan with the sonographer blinded to the AI results. The inter-rater agreement will be determined using Kappa statistics. The results will demonstrate the strength of relationship between the two methods. A strong agreement between the two may facilitate further investigation into the uses of AI, such as use as a teaching tool or in aiding decisions in cases that Sonographers find more difficult to assess such as those patients with a high BMI.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or over
* General Practitioner (GP) and Outpatients (OP) referral
* NAFLD, Unknown, Diabetes, Other metabolic disease

Exclusion Criteria:

* Younger than 18 years old
* Inpatients
* Known large liver masses
* Poor visualisation of the liver due to body type or anatomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be of patients having liver scans or abdominal scans including the liver at Bronglais Hospital, Aberystwyth during the period the study.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Sonographer assessment of the liver | all measurements obtained within single 30 minute appointment
  Sonographers grade the liver normal, mild, moderate, severe fatty liver dependent on factors including hepatorenal contrast, visualisation of vessel borders and of diaphragm.
Measurement of liver fat using attenuation imaging | all measurements obtained within single 30 minute appointment
  Sonographer uses attenuation imaging function to measure liver fd

SECONDARY OUTCOMES:
Age of patient | all measurements obtained within single 30 minute appointment
  Age of patient
Height | all measurements obtained within single 30 minute appointment
  Height, patients height measured immediately after scan.
Weight | all measurements obtained within single 30 minute appointment
  Weight, patient weighed immediately after scan
Diagnosis or Relevant history | all measurements obtained within single 30 minute appointment
  Diagnosis or relevant history from referral form.

CONTACTS AND LOCATIONS:
Locations (1):
- Bronglais Hospital, Aberystwyth, Ceredigion, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT06552377/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT06552377/ICF_001.pdf